CLINICAL TRIAL: NCT04363827
Title: PROTECT: A Randomized Study With Hydroxychloroquine Versus Observational Support for Prevention or Early Phase Treatment of Coronavirus Disease (COVID-19)
Brief Title: Protect: Study With Hydroxychloroquine for Prevention and Early Phase Treatment of Coronavirus Disease (COVID-19)
Acronym: PROTECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting subjects were observed soon after the study was initiated. This difficulty was attributed to the decreased incidence of infections which occurred in the period following the first lock down.
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.47
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: COVID19; Hydroxychloroquine; Prophylaxis; Treatment; SARS-CoV-2
Keywords: COVID19; Households; Hydroxychloroquine; prophylaxis; early phase treatment; prevention; asymptomatic; paucisymptomatic; home situation; SARS-CoV-2-exposed subjects
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Hydroxychloroquine (Experimental): A loading dose Hydroxychloroquine 400 mg twice daily at day 1, followed by a weekly dose of Hydroxychloroquine 200 mg twice daily on days 8, 15 and 22, covering a total of 1 month of treatment.
  Interventions: Drug: Hydroxychloroquine
- Group 1: Observation (No Intervention): observation only
- Group 2: Hydroxycloroquine (Experimental): A loading dose Hydroxychloroquine 400 mg twice daily at day 1 followed by 200 mg twice daily for a total of at least 5-7 days according to clinical evolution.
  Interventions: Drug: Hydroxychloroquine
- Group 2: Observation (No Intervention): Observation only

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine
  Arms: Group 1: Hydroxychloroquine; Group 2: Hydroxycloroquine

SUMMARY:
This is a Italian, superiority, open label cluster-randomised, interventional clinical trial aimed at assessing whether the treatment with Hydroxychloroquine can reduce the percentage of symptomatic subjects compared to observation only in household members/contacts of COVID-19 patients (Group 1) and if the treatment with Hydroxychloroquine could be introduced in early phase COVID-19 population (Group 2).

The participants will be randomised to receive either:

Arm A) hydroxychloroquine vs Arm B) Observation (2:1 randomisation).

DETAILED DESCRIPTION:
This is an open label, superiority, cluster-randomized Italian interventional clinical trial, evaluating the role of Hydroxychloroquine versus observation only in preventing infection to COVID-19 or treating early phase COVID-19 patients.

Each index case is randomised to either Arm A: Hydroxychloroquine or Arm B: observation in a 2:1 ratio on an open label basis. Participants in the same cluster receive the same intervention.

Study population is constituted by:

Group 1: Severe Acute Respiratory Syndrome (SARS) - Corona Virus (CoV)-2-exposed subjects , as household members/contacts of COVID-19 patients.

Group 2: Patients with COVID-19 asymptomatic or paucisymptomatic in home situation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged >= 18 years
2. SARS-CoV-2-exposed subjects, as household members and/or contacts of COVID-19 patients (Group 1). In this group are included Health care professionals in contact with COVID-19 patients.

   or
3. COVID-19 patients, asymptomatic or paucisymptomatic in home situation who are not in treatment with any anti COVID-19 medication (Group 2)
4. Absence of any COVID-19 symptom in last week before randomization (fever >37.5°C, cough, dyspnea) (only for group 1 subjects)
5. Paracetamol treatment is accepted only for group 2.
6. Participant is willing and able to give informed consent for participation in the study (either recorded during a telephonic interview or signed in person) and agrees with the study and its conduct.

Exclusion Criteria:

1. Reported anamnesis for:

   1. Intolerance or previous toxicity for hydroxychloroquine/chloroquine
   2. Bradycardia or reduction rhythm of heart with arrythmias
   3. Ischemic heart disease
   4. Retinopathy
   5. Congestive heart failure under/with use of diuretics
   6. Favism or glucose-6-phosphate dehydrogenase (G6PD) deficiency
   7. Diabetes type 1
   8. Major comorbidities like advanced chronic kidney disease or dialysis therapy, known history of ventricular arrhythmias, any oncologic/hematologic malignancy.
   9. Severe neurological and mental illness
2. Any other contraindication to take hydroxychloroquine
3. Already taking chloroquine, hydroxychloroquine or analogous during the past 3 weeks
4. Use of other antiviral agents in the last 3 weeks
5. Subject with a positive test for SARS-CoV-2 (for Group 1)
6. Pregnant or lactating
7. Current use of medications with known significant drug-drug interactions: digoxin, hypoglycemic agents, anticonvulsant, Cyclosporine, Phenylbutazone, drugs that inhibit CYP2D6
8. Known prolonged QT syndrome or current use of drugs with known QT prolongation
9. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects of Group 1 who become symptomatic and/or swab positive in each arm within 1 month from randomization. | within 1 month from randomization
  Group 1:The primary endpoint/outcome measure is the proportion of subjects of Group 1 who become symptomatic and/or swab positive in each arm within 1 month from randomization.
the proportion of subjects of Group 2 who become swab negative in each arm within 14 days from randomization. | within 14 days from randomization
  Group 2: The primary endpoint/outcome measure is the proportion of subjects of Group 2 who become swab negative in each arm within 14 days from randomization.

SECONDARY OUTCOMES:
The proportion of subjects with positive swabs in Group 1 within 1 month from randomization in both arms | within 1 month from randomization
  The proportion of subjects with positive swabs in randomized population of SARS-CoV-2-exposed subjects ( Group 1) within 1 month from randomization in both arms
The proportion of subjects of Group 1 who become symptomatic in each arm within 1 month from randomization | within 1 month from randomization
  The proportion of subjects of Group 1 who become symptomatic in each arm within 1 month from randomization, in subgroup population identified by stratification factors, class of age and gender.
The proportion of subjects of Group 2 who become swab negative in each arm within 14 days from randomization. | within 14 days from randomization
  The proportion of subjects of Group 2 who become swab negative in each arm within 14 days from randomization, in subgroup population identified by stratification factors, class of age and gender.
The proportion of subjects of Group 2 who become swab negative in each arm within 1 month from randomization in overall population and in subgroup population | within 1 month from randomization
  The proportion of subjects of Group 2 who become swab negative in each arm within 1 month from randomization in overall population and in subgroup population identified by stratification factors, class of age and gender.
Absolute and relative frequencies of Serious Adverse Events | up to 10 months
  Absolute and relative frequencies of Serious Adverse Events (CTCAE version 5.0) in both arms for the Group 1 and Group 2.
Variation in Quality of Life scores in different time points | up to 10 months
  Variation in Quality of Life scores EQ-5D-5L (EQ-5D descriptive system with 5 severity levels from better to worse, and the EQ visual analogue scale (EQ VAS, scale from 100 to 0, high is better) in different time points (weekly) respect to baseline values in both Group 1 and Group 2 populations.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Prof., Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST IRCCS , Meldola Italy; Pierluigi Viale, Prof., Study Chair — Univeristy of Bologna
Locations (1):
- Irst Irccs, Meldola, FC, Italy

REFERENCES:
- [Derived] Nanni O, Viale P, Vertogen B, Lilli C, Zingaretti C, Donati C, Masini C, Monti M, Serra P, Vespignani R, Grossi V, Biggeri A, Scarpi E, Galardi F, Bertoni L, Colamartini A, Falcini F, Altini M, Massa I, Gaggeri R, Martinelli G. PROTECT Trial: A cluster-randomized study with hydroxychloroquine versus observational support for prevention or early-phase treatment of Coronavirus disease (COVID-19): A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Jul 31;21(1):689. doi: 10.1186/s13063-020-04527-4. PMID 32736597